CLINICAL TRIAL: NCT00755729
Title: The Effect of the Preoperative Oral Carbohydrate Attenuating Immediate Postoperative Insulin Resistance on PI3K Dependent Signaling Pathway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Qiang Wang, MD, Shanghai Chang Zheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SCZH-0809-110
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Colorectal Disease
Keywords: Preoperative oral carbohydrate; Insulin resistance; phosphatidylinositol-3-kinase
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCH (Experimental): fast from midnight the night before surgery, and consume 400 ml Nutricia preOp® (12.5% carbohydrates, 0.5 kcal/ml, 240 mOsm, pH 4.9, Nutricia Zoetermeer, The Netherlands) 3 hours prior to induction of anaesthesia and finished the ingestion within 1 hour
  Interventions: Dietary Supplement: Preoperative Oral Carbohydrate
- FSD (No Intervention): fast from midnight the night before surgery, and no preoperative oral carbohydrate loading
  Interventions: Dietary Supplement: Preoperative Oral Carbohydrate

INTERVENTIONS:
Dietary Supplement: Preoperative Oral Carbohydrate — Patients in OCH group consumed 400 ml Nutricia preOp® (12.5% carbohydrates, 0.5 kcal/ml, 240 mOsm, pH 4.9, Nutricia Zoetermeer, The Netherlands) 3 hours prior to induction of anaesthesia and finished the ingestion within 1 hour
  Arms: OCH
Dietary Supplement: Preoperative Oral Carbohydrate — Patients in FSD group were fasted from midnight the night before surgery, and no preoperative oral carbohydrate loading
  Arms: FSD

SUMMARY:
The purpose of this study is to delineate the effects of preoperative oral carbohydrate on immediate postoperative insulin resistance (PIR) in patients undergoing elective open colorectal cancer resection, and to further clarify the hypotheses that preoperative oral carbohydrate treatment attenuates PIR in patients by enhancing insulin signaling to PI3K-dependent pathway.

DETAILED DESCRIPTION:
Postoperative insulin resistance (PIR) is a central feature of postoperative metabolism response to surgical injury, resulting in decreased insulin-stimulated glucose uptake in skeletal muscle and adipose tissue, increased glucose release and hyperglycaemia. The PIR is most pronounced on the day after surgery and lasts for about 3 weeks after uncomplicated elective open abdominal operations, and has been considered as a factor of clinical importance for the postoperative patient. Recent evidences have elucidated the toxicity of hyperglycemia and suggest a causal relation between PIR and complications in the postoperative state and the degree of PIR has been considered as an independent factor determining the length of postoperative hospital stay.

The degree of PIR is proportional to the degree of surgical trauma. Although overcoming PIR by insulin infusion is one way of combating hyperglycemia, prevention of its development can also be achieved by preoperative oral carbohydrate instead of overnight fasting which proven in different kinds of surgery, such as in total hip replacement surgery, colorectal surgery and in elderly patients undergoing coronary artery bypass grafting. As a single intervention in patients given 2-3 hours before anaesthesia, the efficacy of preoperative oral carbohydrate has been shown to be equally as good as the intravenous infusion of glucose with regard to PIR, and attenuated the development of PIR by 50% measured on the first postoperative day after major abdominal surgery. In a placebo-controlled randomized controlled trial of 65 patients undergoing major abdominal surgery, patients who received preoperative oral carbohydrate lost 0.5 cm of the mid-arm circumference by discharge, while the placebo group had more than twice the reduction (1.1 cm). Furthermore, patients receiving the oral carbohydrate-rich beverage before colorectal surgery had a smaller reduction in their quadriceps muscle strength after the operation up to 1 month than those without carbohydrate-rich beverage. These studies suggest that whole-body protein balance, muscle function as well as the suppressive effect of insulin on endogenous glucose release are better maintained and enhanced when patients receive a carbohydrate-rich beverage before surgery. Moreover, in patients who undergo surgery of moderate to severe degree of PIR, the PIR can be overcome if a sufficient amount of insulin is infused to maintain euglycemia, and both glucose uptake and whole body substrate utilization could be normalized in the presence of elevated insulin concentrations. The intensive insulin treatment to maintain normoglycaemia in post-surgical patients in intensive care unit substantially reduces morbidity and mortality. These findings show that excessive insulin can compensate for the defects in insulin action as well, suggesting that PIR might be due to a block in intracellular mechanisms that lead to the decrease in glucose uptake.

The human insulin receptor is a transmembrane glycoprotein, whose cytoplasmic domain contains an insulin-activated protein tyrosine kinase (PTK). Insulin signaling is initiated by binding of insulin to the extracellular α-subunit of insulin receptor, resulting in the stimulation of β-subunit, which contains intrinsic receptor tyrosine kinase activity, autophosphorylation of the receptor at multiple tyrosine residues. Autophosphorylation of the receptor enhances the intrinsic tyrosine kinase activity and evokes a series of phosphorylation events. These include tyrosyl phosphorylation of intracellular substrates named insulin receptor substrates (IRS 1 to 4), phosphatidylinositol-3-kinase (PI3K), and protein kinase B (PKB). The phosphorylated proteins mediate the cellular actions of insulin. On the other hand, the glucose uptake stimulated by insulin in muscle and adipocytes is through the translocation of glucose transporters 4 (GLUT4) from intracellular pools to the plasma membrane. The translocation of GLUT4 to plasma membrane was established to be mediated by PI3K, based on the use of pharmacological inhibitors and expression of a dominant negative mutant or constitutively active form of PI3K.

As molecular switch to regulate the activity of serine/threonine-specifc kinase, PTK and PI3K signaling pathways act cascades important in mediating insulin's effects on endpoint responses. Defects in the receptor kinase activity and signal transduction in the skeletal muscle have been shown previously as a major contributor to the pathogenesis of insulin-resistant states, such as obesity and type II diabetes. Despite these findings, the mechanism by which preoperative oral carbohydrate beverage consumption exerts the effect that attenuating immediate PIR in patients is still unknown. Defects of insulin signal transduction via PI3K-dependent pathway may be possible involved in the development of PIR, and are highly speculated as the main molecular signaling mechanism.

ELIGIBILITY:
Inclusion Criteria:

* The present study employed 32 patients, who underwent elective open colorectal resection for colorectal carcinoma

Exclusion Criteria:

* Diabetes mellitus or impaired glucose tolerance
* Medication affecting insulin sensitivity
* Weight loss greater than 10 per cent during the previous 6 months
* Signs of distant metastasis by CT scanning
* Renal insufficiency (creatinine, > 3 mg/dl; hemodialysis)
* Hepatic insufficiency (Child-Pugh class, ≥ B)
* Gastro-oesophageal reflux disease
* Gastrointestinal obstruction
* Conditions (including pharmacological treatment) known to affect gastric emptying rate

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
PTK activity and PI3K, PKB, GLUT4 expression in rectus abdominis muscle samples by the end of operation | 1 month (postoperative period)

SECONDARY OUTCOMES:
Preoperative general well-beings and the insulin resistance before and immediately after surgery assessed with the visual analogue scale (VAS) and the homeostasis model assessment (HOMA) respectively | Perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD, Study Chair — Shanghai Chang Zheng Hospital; Zhi Guo Wang, MD, Principal Investigator — Department of General Surgery, Shanghai Chang Zheng Hospital
Locations (1):
- Department of General Surgery, Shanghai Chang Zheng Hospital,, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang ZG, Wang Q, Wang WJ, Qin HL. Randomized clinical trial to compare the effects of preoperative oral carbohydrate versus placebo on insulin resistance after colorectal surgery. Br J Surg. 2010 Mar;97(3):317-27. doi: 10.1002/bjs.6963. PMID 20101593